CLINICAL TRIAL: NCT02177318
Title: Drug Use Results Survey of Tiotropium Bromide
Brief Title: Tiotropium in the Treatment of the Patients With Chronic Obstructive Pulmonary Disease
Acronym: COPD
Status: Completed | Type: Observational
Sponsor: Boehringer Ingelheim (Industry)
Responsible Party: Sponsor
Other Study IDs: 205.314
Record Dates: First submitted 2008-01-31; First posted 2014-06-27 (Estimated); Last update posted 2014-06-27 (Estimated); Status verified 2014-06

CONDITIONS: Pulmonary Disease, Chronic Obstructive
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive | interventions — Tiotropium Bromide; Inhalation

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective

GROUPS / COHORTS (1):
- Patients with COPD
  Interventions: Drug: Spiriva (tiotropium bromide) inhalation capsules

INTERVENTIONS:
Drug: Spiriva (tiotropium bromide) inhalation capsules — Survey of patients with COPD using Spiriva (tiotropium bromide) inhalation capsules

SUMMARY:
To collect post-marketing safety and effectiveness information on the use of Tiotropium Inhalation Capsules (18 μg) in patients with chronic obstructive pulmonary disease in daily clinical settings

ELIGIBILITY:
Inclusion Criteria:

- Patients with COPD

Exclusion Criteria:

-There is no exclusion criterion, because this post marketing study (PMS) is observational survey under condition of normal clinical practice

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: COPD patients in daily clinical settings.
Sampling Method: Non-Probability Sample
Enrollment: 3588 (Actual)
Dates: Start 2005-04; Primary Completion 2007-09 (Actual)

PRIMARY OUTCOMES:
Number of patients with adverse events | Up to 4 weeks after start of treatment
Number of patients with adverse drug reactions | Up to 4 weeks after start of treatment
Number of patients with serious adverse events | Up to 4 weeks after start of treatment

SECONDARY OUTCOMES:
Physician's overall judgement by medical interview into four grades: 1. Improved 2. No Change 3. Aggravated 4.Unassessable | Up to 4 weeks after start of treatment

CONTACTS AND LOCATIONS:
Overall Officials: Boehringer Ingelheim, Study Chair — Boehringer Ingelheim
Locations (416):
- Japan (416):
  - Boehringer Ingelheim Investigational Site, Abashiri
  - Boehringer Ingelheim Investigational Site, Aizu-Wakamatsu
  - Boehringer Ingelheim Investigational Site, Aizubangemachi
  - Boehringer Ingelheim Investigational Site, Aizumisatomachi
  - Boehringer Ingelheim Investigational Site, Akashi
  - Boehringer Ingelheim Investigational Site, Akita
  - Boehringer Ingelheim Investigational Site, Akō
  - Boehringer Ingelheim Investigational Site, Amagasaki
  - Boehringer Ingelheim Investigational Site, Amakusa
  - Boehringer Ingelheim Investigational Site, Amimachi
  - Boehringer Ingelheim Investigational Site, Anan
  - Boehringer Ingelheim Investigational Site, Anjo
  - Boehringer Ingelheim Investigational Site, Arakawamachi
  - Boehringer Ingelheim Investigational Site, Arao
  - Boehringer Ingelheim Investigational Site, Aritacho
  - Boehringer Ingelheim Investigational Site, Asahikawa
  - Boehringer Ingelheim Investigational Site, Ashikaga
  - Boehringer Ingelheim Investigational Site, Atami
  - Boehringer Ingelheim Investigational Site, Atsugi
  - Boehringer Ingelheim Investigational Site, Awa
  - Boehringer Ingelheim Investigational Site, Ayabe
  - Boehringer Ingelheim Investigational Site, Ayagawacho
  - Boehringer Ingelheim Investigational Site, Ayase
  - Boehringer Ingelheim Investigational Site, Beppu
  - Boehringer Ingelheim Investigational Site, Bibai
  - Boehringer Ingelheim Investigational Site, Bungoohno
  - Boehringer Ingelheim Investigational Site, Chiba
  - Boehringer Ingelheim Investigational Site, Chigasaki
  - Boehringer Ingelheim Investigational Site, Chikusei
  - Boehringer Ingelheim Investigational Site, Chikushino-shi
  - Boehringer Ingelheim Investigational Site, Chitose
  - Boehringer Ingelheim Investigational Site, Date
  - Boehringer Ingelheim Investigational Site, Ebetsu
  - Boehringer Ingelheim Investigational Site, Echizen
  - Boehringer Ingelheim Investigational Site, Emukaecho
  - Boehringer Ingelheim Investigational Site, Engarucho
  - Boehringer Ingelheim Investigational Site, Fuchū
  - Boehringer Ingelheim Investigational Site, Fuji
  - Boehringer Ingelheim Investigational Site, Fujiidera
  - Boehringer Ingelheim Investigational Site, Fujikawaguchiko
  - Boehringer Ingelheim Investigational Site, Fujinomiya
  - Boehringer Ingelheim Investigational Site, Fukagawa
  - Boehringer Ingelheim Investigational Site, Fukaya
  - Boehringer Ingelheim Investigational Site, Fukuchiyama
  - Boehringer Ingelheim Investigational Site, Fukui
  - Boehringer Ingelheim Investigational Site, Fukuoka
  - Boehringer Ingelheim Investigational Site, Fukuroi
  - Boehringer Ingelheim Investigational Site, Fukushima
  - Boehringer Ingelheim Investigational Site, Fukutsu
  - Boehringer Ingelheim Investigational Site, Fukuyama
  - Boehringer Ingelheim Investigational Site, Funabashi
  - Boehringer Ingelheim Investigational Site, Futabamachi
  - Boehringer Ingelheim Investigational Site, Geiseimura
  - Boehringer Ingelheim Investigational Site, Gifu
  - Boehringer Ingelheim Investigational Site, Ginowan
  - Boehringer Ingelheim Investigational Site, Gobō
  - Boehringer Ingelheim Investigational Site, Gosen
  - Boehringer Ingelheim Investigational Site, Gotemba
  - Boehringer Ingelheim Investigational Site, Gyouda
  - Boehringer Ingelheim Investigational Site, Habikino
  - Boehringer Ingelheim Investigational Site, Hachinohe
  - Boehringer Ingelheim Investigational Site, Hachirogatamachi
  - Boehringer Ingelheim Investigational Site, Hagi
  - Boehringer Ingelheim Investigational Site, Hakodate
  - Boehringer Ingelheim Investigational Site, Hakusan
  - Boehringer Ingelheim Investigational Site, Hamada
  - Boehringer Ingelheim Investigational Site, Hamamatsu
  - Boehringer Ingelheim Investigational Site, Handa
  - Boehringer Ingelheim Investigational Site, Hanyū
  - Boehringer Ingelheim Investigational Site, Hatsukaichi
  - Boehringer Ingelheim Investigational Site, Hayashimacho
  - Boehringer Ingelheim Investigational Site, Higashihiroshima
  - Boehringer Ingelheim Investigational Site, Higashimatsushima
  - Boehringer Ingelheim Investigational Site, Higashiosaka
  - Boehringer Ingelheim Investigational Site, Higashiōmi
  - Boehringer Ingelheim Investigational Site, Hikari
  - Boehringer Ingelheim Investigational Site, Himeji
  - Boehringer Ingelheim Investigational Site, Hirakata
  - Boehringer Ingelheim Investigational Site, Hiratsuka
  - Boehringer Ingelheim Investigational Site, Hirosaki
  - Boehringer Ingelheim Investigational Site, Hiroshima
  - Boehringer Ingelheim Investigational Site, Hita
  - Boehringer Ingelheim Investigational Site, Hitachi
  - Boehringer Ingelheim Investigational Site, Hitoyoshi
  - Boehringer Ingelheim Investigational Site, Hōfu
  - Boehringer Ingelheim Investigational Site, Iamabari
  - Boehringer Ingelheim Investigational Site, Ibaraki
  - Boehringer Ingelheim Investigational Site, Ibarakimachi
  - Boehringer Ingelheim Investigational Site, Ibigawacho
  - Boehringer Ingelheim Investigational Site, Ibusuki
  - Boehringer Ingelheim Investigational Site, Ichihara
  - Boehringer Ingelheim Investigational Site, Ichinomiya
  - Boehringer Ingelheim Investigational Site, Ichinoseki
  - Boehringer Ingelheim Investigational Site, Iga
  - Boehringer Ingelheim Investigational Site, Iida
  - Boehringer Ingelheim Investigational Site, Iizuka
  - Boehringer Ingelheim Investigational Site, Ikoma
  - Boehringer Ingelheim Investigational Site, Imari
  - Boehringer Ingelheim Investigational Site, Imizu
  - Boehringer Ingelheim Investigational Site, Ina
  - Boehringer Ingelheim Investigational Site, Inazawa
  - Boehringer Ingelheim Investigational Site, Inuyama
  - Boehringer Ingelheim Investigational Site, Isahaya
  - Boehringer Ingelheim Investigational Site, Ise
  - Boehringer Ingelheim Investigational Site, Isehara
  - Boehringer Ingelheim Investigational Site, Ishikari
  - Boehringer Ingelheim Investigational Site, Ishinomaki
  - Boehringer Ingelheim Investigational Site, Itami
  - Boehringer Ingelheim Investigational Site, Itanocho
  - Boehringer Ingelheim Investigational Site, Itō
  - Boehringer Ingelheim Investigational Site, Iwaki
  - Boehringer Ingelheim Investigational Site, Iwakuni
  - Boehringer Ingelheim Investigational Site, Iwamizawa
  - Boehringer Ingelheim Investigational Site, Iwanaicho
  - Boehringer Ingelheim Investigational Site, Iwata
  - Boehringer Ingelheim Investigational Site, Iyo
  - Boehringer Ingelheim Investigational Site, Izu
  - Boehringer Ingelheim Investigational Site, Izumisano
  - Boehringer Ingelheim Investigational Site, Izumo
  - Boehringer Ingelheim Investigational Site, Izunokuni
  - Boehringer Ingelheim Investigational Site, Jimokujicho
  - Boehringer Ingelheim Investigational Site, Jouetsu
  - Boehringer Ingelheim Investigational Site, Jōsō
  - Boehringer Ingelheim Investigational Site, Jōyō
  - Boehringer Ingelheim Investigational Site, Kaga
  - Boehringer Ingelheim Investigational Site, Kagoshima
  - Boehringer Ingelheim Investigational Site, Kaizuka
  - Boehringer Ingelheim Investigational Site, Kajikicho
  - Boehringer Ingelheim Investigational Site, Kakegawa
  - Boehringer Ingelheim Investigational Site, Kami
  - Boehringer Ingelheim Investigational Site, Kamiamakusa
  - Boehringer Ingelheim Investigational Site, Kamisu
  - Boehringer Ingelheim Investigational Site, Kanazawa
  - Boehringer Ingelheim Investigational Site, Kandamachi
  - Boehringer Ingelheim Investigational Site, Kan’onjichō
  - Boehringer Ingelheim Investigational Site, Kasai
  - Boehringer Ingelheim Investigational Site, Kasama
  - Boehringer Ingelheim Investigational Site, Kasaoka
  - Boehringer Ingelheim Investigational Site, Kashihara
  - Boehringer Ingelheim Investigational Site, Kashima
  - Boehringer Ingelheim Investigational Site, Kashiwazaki
  - Boehringer Ingelheim Investigational Site, Kasuga
  - Boehringer Ingelheim Investigational Site, Kasuigai
  - Boehringer Ingelheim Investigational Site, Kasukabe
  - Boehringer Ingelheim Investigational Site, Kasuyamachi
  - Boehringer Ingelheim Investigational Site, Katō
  - Boehringer Ingelheim Investigational Site, Katsuyama
  - Boehringer Ingelheim Investigational Site, Kawachi-Nagano
  - Boehringer Ingelheim Investigational Site, Kawagoe
  - Boehringer Ingelheim Investigational Site, Kawaguchi
  - Boehringer Ingelheim Investigational Site, Kawanishimachi
  - Boehringer Ingelheim Investigational Site, Kawasaki
  - Boehringer Ingelheim Investigational Site, Kayano
  - Boehringer Ingelheim Investigational Site, Kazuno
  - Boehringer Ingelheim Investigational Site, Kinkōchō
  - Boehringer Ingelheim Investigational Site, Kitakami
  - Boehringer Ingelheim Investigational Site, Kitakyushu
  - Boehringer Ingelheim Investigational Site, Kitami
  - Boehringer Ingelheim Investigational Site, Kobe
  - Boehringer Ingelheim Investigational Site, Kochi
  - Boehringer Ingelheim Investigational Site, Koga
  - Boehringer Ingelheim Investigational Site, Komonocho
  - Boehringer Ingelheim Investigational Site, Kouriyama
  - Boehringer Ingelheim Investigational Site, Koushu
  - Boehringer Ingelheim Investigational Site, Kozakaichō
  - Boehringer Ingelheim Investigational Site, Kōnan
  - Boehringer Ingelheim Investigational Site, Kōriyama
  - Boehringer Ingelheim Investigational Site, Kōshi
  - Boehringer Ingelheim Investigational Site, Kudamatsu
  - Boehringer Ingelheim Investigational Site, Kumamoto
  - Boehringer Ingelheim Investigational Site, Kunimimachi
  - Boehringer Ingelheim Investigational Site, Kunisaki
  - Boehringer Ingelheim Investigational Site, Kurashiki
  - Boehringer Ingelheim Investigational Site, Kurayoshi
  - Boehringer Ingelheim Investigational Site, Kure
  - Boehringer Ingelheim Investigational Site, Kurihara
  - Boehringer Ingelheim Investigational Site, Kurume
  - Boehringer Ingelheim Investigational Site, Kushiro
  - Boehringer Ingelheim Investigational Site, Kuwana
  - Boehringer Ingelheim Investigational Site, Kyoto
  - Boehringer Ingelheim Investigational Site, Kyōtango
  - Boehringer Ingelheim Investigational Site, Maebashi
  - Boehringer Ingelheim Investigational Site, Marugame
  - Boehringer Ingelheim Investigational Site, Masuda
  - Boehringer Ingelheim Investigational Site, Matsudo
  - Boehringer Ingelheim Investigational Site, Matsue
  - Boehringer Ingelheim Investigational Site, Matsumoto
  - Boehringer Ingelheim Investigational Site, Matsusaka
  - Boehringer Ingelheim Investigational Site, Matsuyama
  - Boehringer Ingelheim Investigational Site, Mibumachi
  - Boehringer Ingelheim Investigational Site, Mihamacho
  - Boehringer Ingelheim Investigational Site, Mihara
  - Boehringer Ingelheim Investigational Site, Minamisatsuma
  - Boehringer Ingelheim Investigational Site, Minamisouma
  - Boehringer Ingelheim Investigational Site, Minamiuonuma
  - Boehringer Ingelheim Investigational Site, Mino
  - Boehringer Ingelheim Investigational Site, Minoh
  - Boehringer Ingelheim Investigational Site, Misasacho
  - Boehringer Ingelheim Investigational Site, Misato
  - Boehringer Ingelheim Investigational Site, Mishima
  - Boehringer Ingelheim Investigational Site, Mito
  - Boehringer Ingelheim Investigational Site, Miyakicho
  - Boehringer Ingelheim Investigational Site, Miyakonojō
  - Boehringer Ingelheim Investigational Site, Miyazaki
  - Boehringer Ingelheim Investigational Site, Miyoshi
  - Boehringer Ingelheim Investigational Site, Mizunami
  - Boehringer Ingelheim Investigational Site, Mobara
  - Boehringer Ingelheim Investigational Site, Moriguchi
  - Boehringer Ingelheim Investigational Site, Morioka
  - Boehringer Ingelheim Investigational Site, Muroran
  - Boehringer Ingelheim Investigational Site, Nabari
  - Boehringer Ingelheim Investigational Site, Nagahama
  - Boehringer Ingelheim Investigational Site, Nagano
  - Boehringer Ingelheim Investigational Site, Nagaoka
  - Boehringer Ingelheim Investigational Site, Nagasaki
  - Boehringer Ingelheim Investigational Site, Nagato
  - Boehringer Ingelheim Investigational Site, Nago
  - Boehringer Ingelheim Investigational Site, Nagoya
  - Boehringer Ingelheim Investigational Site, Naha
  - Boehringer Ingelheim Investigational Site, Nakama
  - Boehringer Ingelheim Investigational Site, Nakashibetsucho
  - Boehringer Ingelheim Investigational Site, Nanao
  - Boehringer Ingelheim Investigational Site, Nankoku
  - Boehringer Ingelheim Investigational Site, Nantan
  - Boehringer Ingelheim Investigational Site, Nara
  - Boehringer Ingelheim Investigational Site, Narutō
  - Boehringer Ingelheim Investigational Site, Nasukarasuyama
  - Boehringer Ingelheim Investigational Site, Neyagawa
  - Boehringer Ingelheim Investigational Site, Nihonmatsu
  - Boehringer Ingelheim Investigational Site, Niigata
  - Boehringer Ingelheim Investigational Site, Niihamashi
  - Boehringer Ingelheim Investigational Site, Nikkō
  - Boehringer Ingelheim Investigational Site, Nishiiyo
  - Boehringer Ingelheim Investigational Site, Nishinomiya
  - Boehringer Ingelheim Investigational Site, Nishio
  - Boehringer Ingelheim Investigational Site, Nobeoka
  - Boehringer Ingelheim Investigational Site, Noboribetsu
  - Boehringer Ingelheim Investigational Site, Noda
  - Boehringer Ingelheim Investigational Site, Nomi
  - Boehringer Ingelheim Investigational Site, Noshiro
  - Boehringer Ingelheim Investigational Site, Notōchō
  - Boehringer Ingelheim Investigational Site, Numata
  - Boehringer Ingelheim Investigational Site, Numazu
  - Boehringer Ingelheim Investigational Site, Oaraimachi
  - Boehringer Ingelheim Investigational Site, Obama
  - Boehringer Ingelheim Investigational Site, Obihiro
  - Boehringer Ingelheim Investigational Site, Odawara
  - Boehringer Ingelheim Investigational Site, Ogawaramachi
  - Boehringer Ingelheim Investigational Site, Ogi
  - Boehringer Ingelheim Investigational Site, Ojiya
  - Boehringer Ingelheim Investigational Site, Okayama
  - Boehringer Ingelheim Investigational Site, Okinawa
  - Boehringer Ingelheim Investigational Site, Omuta
  - Boehringer Ingelheim Investigational Site, Osaka
  - Boehringer Ingelheim Investigational Site, Otaru
  - Boehringer Ingelheim Investigational Site, Owariasahi
  - Boehringer Ingelheim Investigational Site, Ōdate
  - Boehringer Ingelheim Investigational Site, Ōita
  - Boehringer Ingelheim Investigational Site, Ōmihachiman
  - Boehringer Ingelheim Investigational Site, Ōnomachi
  - Boehringer Ingelheim Investigational Site, Ōta-ku
  - Boehringer Ingelheim Investigational Site, Ōtake
  - Boehringer Ingelheim Investigational Site, Ōtsu
  - Boehringer Ingelheim Investigational Site, Ōtsumachi
  - Boehringer Ingelheim Investigational Site, Rittō
  - Boehringer Ingelheim Investigational Site, Ryūgasaki
  - Boehringer Ingelheim Investigational Site, Sado
  - Boehringer Ingelheim Investigational Site, Saga
  - Boehringer Ingelheim Investigational Site, Sagamihara
  - Boehringer Ingelheim Investigational Site, Saiki
  - Boehringer Ingelheim Investigational Site, Saitama
  - Boehringer Ingelheim Investigational Site, Sakacho
  - Boehringer Ingelheim Investigational Site, Sakai
  - Boehringer Ingelheim Investigational Site, Sakaimachi
  - Boehringer Ingelheim Investigational Site, Sakaiminato
  - Boehringer Ingelheim Investigational Site, Sakata
  - Boehringer Ingelheim Investigational Site, Saku
  - Boehringer Ingelheim Investigational Site, Sanjyo
  - Boehringer Ingelheim Investigational Site, Sanuki
  - Boehringer Ingelheim Investigational Site, Sanyōonoda
  - Boehringer Ingelheim Investigational Site, Sapporo
  - Boehringer Ingelheim Investigational Site, Sasayama
  - Boehringer Ingelheim Investigational Site, Sasebo
  - Boehringer Ingelheim Investigational Site, Sayama
  - Boehringer Ingelheim Investigational Site, Sendai
  - Boehringer Ingelheim Investigational Site, Sennan
  - Boehringer Ingelheim Investigational Site, Shibetsu
  - Boehringer Ingelheim Investigational Site, Shibukawa
  - Boehringer Ingelheim Investigational Site, Shimada
  - Boehringer Ingelheim Investigational Site, Shimonoseki
  - Boehringer Ingelheim Investigational Site, Shimotsuke
  - Boehringer Ingelheim Investigational Site, Shimotsuma
  - Boehringer Ingelheim Investigational Site, Shingū
  - Boehringer Ingelheim Investigational Site, Shiogama
  - Boehringer Ingelheim Investigational Site, Shirahamachō
  - Boehringer Ingelheim Investigational Site, Shiroishi
  - Boehringer Ingelheim Investigational Site, Shiroishichō
  - Boehringer Ingelheim Investigational Site, Shizuoka
  - Boehringer Ingelheim Investigational Site, Shoocho
  - Boehringer Ingelheim Investigational Site, Shūnan
  - Boehringer Ingelheim Investigational Site, Soo
  - Boehringer Ingelheim Investigational Site, Souka
  - Boehringer Ingelheim Investigational Site, Suita
  - Boehringer Ingelheim Investigational Site, Sukagawa
  - Boehringer Ingelheim Investigational Site, Sukumo
  - Boehringer Ingelheim Investigational Site, Sunagawa
  - Boehringer Ingelheim Investigational Site, Susono
  - Boehringer Ingelheim Investigational Site, Suwa
  - Boehringer Ingelheim Investigational Site, Suzuka
  - Boehringer Ingelheim Investigational Site, Tagawa
  - Boehringer Ingelheim Investigational Site, Tainai
  - Boehringer Ingelheim Investigational Site, Takahashi
  - Boehringer Ingelheim Investigational Site, Takamatsu
  - Boehringer Ingelheim Investigational Site, Takaoka
  - Boehringer Ingelheim Investigational Site, Takarazuka
  - Boehringer Ingelheim Investigational Site, Takasago
  - Boehringer Ingelheim Investigational Site, Takashima
  - Boehringer Ingelheim Investigational Site, Takatsuki
  - Boehringer Ingelheim Investigational Site, Taku
  - Boehringer Ingelheim Investigational Site, Tamana
  - Boehringer Ingelheim Investigational Site, Tamano
  - Boehringer Ingelheim Investigational Site, Tanabe
  - Boehringer Ingelheim Investigational Site, Taragimachi
  - Boehringer Ingelheim Investigational Site, Tenri
  - Boehringer Ingelheim Investigational Site, Tokaimura
  - Boehringer Ingelheim Investigational Site, Tokorozawa
  - Boehringer Ingelheim Investigational Site, Tokunoshimacho
  - Boehringer Ingelheim Investigational Site, Tokushima
  - Boehringer Ingelheim Investigational Site, Tokyo Adachi-ku
  - Boehringer Ingelheim Investigational Site, Tokyo Akishima
  - Boehringer Ingelheim Investigational Site, Tokyo Bunkyo-ku
  - Boehringer Ingelheim Investigational Site, Tokyo Chiyoda-ku
  - Boehringer Ingelheim Investigational Site, Tokyo Edogawa-ku
  - Boehringer Ingelheim Investigational Site, Tokyo Hachioji
  - Boehringer Ingelheim Investigational Site, Tokyo Higashimurayama
  - Boehringer Ingelheim Investigational Site, Tokyo Higashiyamato
  - Boehringer Ingelheim Investigational Site, Tokyo Hino
  - Boehringer Ingelheim Investigational Site, Tokyo Itabashi-ku
  - Boehringer Ingelheim Investigational Site, Tokyo Katsushika-ku
  - Boehringer Ingelheim Investigational Site, Tokyo Kiyose
  - Boehringer Ingelheim Investigational Site, Tokyo Komae
  - Boehringer Ingelheim Investigational Site, Tokyo Koto-ku
  - Boehringer Ingelheim Investigational Site, Tokyo Meguro-ku
  - Boehringer Ingelheim Investigational Site, Tokyo Minato-ku
  - Boehringer Ingelheim Investigational Site, Tokyo Nakano-ku
  - Boehringer Ingelheim Investigational Site, Tokyo Nerima-ku
  - Boehringer Ingelheim Investigational Site, Tokyo Nishitokyo
  - Boehringer Ingelheim Investigational Site, Tokyo Ome
  - Boehringer Ingelheim Investigational Site, Tokyo Ota-ku
  - Boehringer Ingelheim Investigational Site, Tokyo Setagaya-ku
  - Boehringer Ingelheim Investigational Site, Tokyo Shibuya-ku
  - Boehringer Ingelheim Investigational Site, Tokyo Shinagawa-ku
  - Boehringer Ingelheim Investigational Site, Tokyo Shinjuku-ku
  - Boehringer Ingelheim Investigational Site, Tokyo Suginami-ku
  - Boehringer Ingelheim Investigational Site, Tokyo Sumida-ku
  - Boehringer Ingelheim Investigational Site, Tokyo Taito-ku
  - Boehringer Ingelheim Investigational Site, Tokyo Toshima-ku
  - Boehringer Ingelheim Investigational Site, Tomakomai
  - Boehringer Ingelheim Investigational Site, Tomigusu
  - Boehringer Ingelheim Investigational Site, Tomioka
  - Boehringer Ingelheim Investigational Site, Tondabayashi
  - Boehringer Ingelheim Investigational Site, Toride
  - Boehringer Ingelheim Investigational Site, Tottori
  - Boehringer Ingelheim Investigational Site, Toyama
  - Boehringer Ingelheim Investigational Site, Toyohashi
  - Boehringer Ingelheim Investigational Site, Toyokawa
  - Boehringer Ingelheim Investigational Site, Toyooka
  - Boehringer Ingelheim Investigational Site, Toyosatocho
  - Boehringer Ingelheim Investigational Site, Toyota
  - Boehringer Ingelheim Investigational Site, Tōkamachi
  - Boehringer Ingelheim Investigational Site, Tsu
  - Boehringer Ingelheim Investigational Site, Tsukuba
  - Boehringer Ingelheim Investigational Site, Tsurugicho
  - Boehringer Ingelheim Investigational Site, Tsuruoka
  - Boehringer Ingelheim Investigational Site, Tsushima
  - Boehringer Ingelheim Investigational Site, Tsuyama
  - Boehringer Ingelheim Investigational Site, Ube
  - Boehringer Ingelheim Investigational Site, Uchikocho
  - Boehringer Ingelheim Investigational Site, Uchinadamachi
  - Boehringer Ingelheim Investigational Site, Uekimachi
  - Boehringer Ingelheim Investigational Site, Uji
  - Boehringer Ingelheim Investigational Site, Uki
  - Boehringer Ingelheim Investigational Site, Unzen
  - Boehringer Ingelheim Investigational Site, Urakawacho
  - Boehringer Ingelheim Investigational Site, Urasoe
  - Boehringer Ingelheim Investigational Site, Urayasu
  - Boehringer Ingelheim Investigational Site, Uruma
  - Boehringer Ingelheim Investigational Site, Usa
  - Boehringer Ingelheim Investigational Site, Usuki
  - Boehringer Ingelheim Investigational Site, Utsunomiya
  - Boehringer Ingelheim Investigational Site, Wakayama
  - Boehringer Ingelheim Investigational Site, Yabu
  - Boehringer Ingelheim Investigational Site, Yachimata
  - Boehringer Ingelheim Investigational Site, Yachiyo
  - Boehringer Ingelheim Investigational Site, Yaizu
  - Boehringer Ingelheim Investigational Site, Yakumochō
  - Boehringer Ingelheim Investigational Site, Yakushimacho
  - Boehringer Ingelheim Investigational Site, Yamaga
  - Boehringer Ingelheim Investigational Site, Yamagata
  - Boehringer Ingelheim Investigational Site, Yamato
  - Boehringer Ingelheim Investigational Site, Yamatotakada
  - Boehringer Ingelheim Investigational Site, Yanai
  - Boehringer Ingelheim Investigational Site, Yao
  - Boehringer Ingelheim Investigational Site, Yatomi
  - Boehringer Ingelheim Investigational Site, Yatsushiro
  - Boehringer Ingelheim Investigational Site, Yawata
  - Boehringer Ingelheim Investigational Site, Yokkaichi
  - Boehringer Ingelheim Investigational Site, Yokohama
  - Boehringer Ingelheim Investigational Site, Yokosuka
  - Boehringer Ingelheim Investigational Site, Yokote
  - Boehringer Ingelheim Investigational Site, Yonabarucho
  - Boehringer Ingelheim Investigational Site, Yonezawa
  - Boehringer Ingelheim Investigational Site, Yorocho
  - Boehringer Ingelheim Investigational Site, Yoshinochō
  - Boehringer Ingelheim Investigational Site, Yufu
  - Boehringer Ingelheim Investigational Site, Yurihonjou